CLINICAL TRIAL: NCT03486366
Title: Application of Novel Diagnostic and Therapeutical Methods in Epilepsy and Neurodevelopmental Abnormalities in Children Based on the Clinical and Cellular Model of the Mammalian Target of Rapamycin - mTOR Dependent Epilepsy.
Brief Title: Application of Novel Diagnostic and Therapeutical Methods in Epilepsy and Neurodevelopmental Abnormalities in Children.
Acronym: EPIMARKER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Children's Memorial Health Institute, Poland (Other)
Responsible Party: Principal Investigator, Sergiusz Jozwiak, Professor Head of Department Neurology in Children Hospital, Medical University of Warsaw
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Strategmed3/306306/4/NCBR/2017
Record Dates: First submitted 2018-03-26; First posted 2018-04-03 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Epilepsy
Keywords: epilepsy, TSC, biomarkers, mTOR pathway
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: With EPIMARKER we aim to develop clinically useful tools enabling accurate and early detection of risk of drug resistant or recurrent seizures and stablish the new therapeutic and preventative possibilities for epilepsy.
  The Epimarker algorithms will include selected data obtained in 3 unique models of epilepsy in developing brain.
  * EEG recordings and clinical data from a prospective study of drug-resistant epilepsy development in young children with TSC,
  * EEG recording and clinical data from a prospective study of epilepsy after antiepileptic drug withdrawal in children with TSC
  * Molecular biomarkers in both above clinical setting, established by means of a broad range of molecular analyses, including a diverse set of cutting edge analyses of blood samples, that will be obtained at study entry, at the onset of drug- resistance or recurrent epilepsy, and after 12-month follow-up and the verified in a Epimarker cellular model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workpackage1 WP1 (Other): Non interventional trial: male or female children with a definite diagnosis of TSC (Roach 1998), aged up to 4 years, diagnosis of epilepsy established on the basis of clinical seizures or epileptiform changes on EEG within 1-7 days prior to baseline. We plan to enroll 60 TSC patients into WP1 to Epimarker in 12 months.
  Interventions: Other: non interventional trial
- Workpackage2 WP2 (Other): Non interventional trial: male or female children with a definite diagnosis of TSC (Roach criteria: Roach 1998) and epilepsy, aged up to 16 years, seizure free, in whom a decision to withdraw antiepileptic drugs was made. We plan to enroll 60 TSC patients into WP2 to Epimarker in 12 months. The data obtained in children seizure free at the end of follow-up and patients with recurrent seizures will be compare.
  Interventions: Other: non interventional trial

INTERVENTIONS:
Other: non interventional trial — other
  Other Names: other

SUMMARY:
Epilepsy affects 1% of the world's population and 6 million people in Europe. The estimated total cost of €20 billion in Europe in 2014 makes epilepsy a significant socioeconomic burden. Despite great progress in the management of epilepsy and increasing numbers of antiepileptic drugs, 30-40% of epilepsy patients are refractory to all available medications. Moreover, in childhood epilepsy is a causative factor of psychiatric and behavioral comorbidities, including developmental delay and autism spectrum disorder. In spite of multiple trials no reliable biomarker of epilepsy development has been identified. There are no studies on biomarkers of drug-resistance or epilepsy recurrence after the drug withdrawal. EPIMARKER is a first project, carried out in humans, which is going to examine in prospective way clinical, electroencephalographic and molecular biomarkers to produce an integrative tool useful in everyday diagnosis and treatment of epilepsy in children to prevent the development of drug-resistant epilepsy and its behavioral comorbidities as mental retardation and autism. The set of molecular biomarkers will be determined by quantitative transcriptomic and proteomic studies and validated in reprogrammed cellular models.

DETAILED DESCRIPTION:
The clinical part of EPIMARKER is composed of 2 prospective studies (WP1 and WP2) of epilepsy progress in Tuberous Sclerosis Complex -TSC children, performed in 2 sites: Medical University of Warsaw -WUM and Children's Memoroal Health Institute - IPCZD, Poland.

WP1 and WP2 are designed to conduct the studies, but the resulting data and samples will be analyzed and used in Workpackage 3-12 (WP3-12).

CLINICAL STUDY in WP1 Inclusion criteria: male or female children with a definite diagnosis of TSC (Roach 1998), aged up to 4 years, diagnosis of epilepsy established on the basis of clinical seizures or epileptiform changes on EEG within 1-7 days prior to baseline , written informed consent of caregivers.

Study overview: Each subject will be followed for 12 month. Epilepsy will be tracked with serial video EEG (vEEG) recordings and clinical investigations performed every 3 months. Apart from medical history of the patients, data from seizure diary, neuroimaging studies, and neuropsychological examinations will be collected. Blood samples for biomarkers studies will be collected at study entry, at the onset of drug- resistant seizures or after 6 months, whichever is applicable, and at the end of follow-up in all patients participating in the project. The data obtained in children responding, to standard and with drug- resistant seizures will be compare.

Sample size: We plan to enroll 60 TSC patients into WP1 of Epimarker in 12 months. Based upon our preliminary results and extensive experience with TSC, we predict that about 50% of patients will develop drug- resistant seizures, while 50% will respond to standard treatment (Jozwiak 2011) Study endpoints: the primary clinical endpoint of this study is a collection of a set of clinical, molecular, and EEG source data in all subjects.

CLINICAL STUDY in WP2 Inclusion criteria: male or female children with a definite diagnosis of TSC (Roach criteria: Roach 1998) and epilepsy, aged up to 16 years, seizure free, in whom a decision to withdraw antiepileptic drugs was made, written informed consent of caregivers.

Study overview: Each subject will be followed for 12 months. Antiepileptic drugs will be withdrawn within 3 months in all subjects starting, at study entry. Epilepsy will be tracked by means of serial video EEG recordings and clinical investigations performed every 3 months. Apart from medical history of the patients, data from seizures diary, neuroimaging studies and neuropsychological examinations will be collected. Patients with recurrent seizures will receive antiepileptic treatment according to current standards. Blood samples for biomarkers study will be collected at study entry, at the end of drugs withdrawal, at the onset recurrent seizures and at the end of follow-up in all patient participating in the project. The data obtained in children seizure free at the end of follow-up and patients with recurrent seizures will be compare.

Sample size: We plan to enroll 60 TSC patients into WP2 of Epimarker in 12 months. Based upon our preliminary results and extensive experience with TSC, we predict that about 50% of patients will develop recurrent seizures, while 50% remain seizure free (unpublished data).

Study endpoints: the primary clinical endpoint of this study is a collection of a set of clinical, molecular, and EEG source data in all subjects.

ELIGIBILITY:
Inclusion Criteria WP1:

* male or female children with a definite diagnosis of TSC (Roach 1998),
* aged up to 4 years,
* diagnosis of epilepsy established on the basis of clinical seizures or
* epileptiform changes on EEG within 1-7 days prior to baseline ,
* written informed consent of caregivers.

Inclusion Criteria WP2:

* male or female children with a definite diagnosis of TSC (Roach criteria: Roach 1998) with epilepsy,
* aged up to 16 years,
* seizure free, in whom a decision to withdraw antiepileptic drugs was made,
* written informed consent of caregivers.

Exclusion Criteria:

-

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
EEG and molecular data collection and integration into clinically applicable tool | 2020
  The EEG algorithm will include the data from automatic statistical analysis of prospectively recorded EEG signal and comprehensive clinical investigations. To achieve this goal, a special automatic system to detect and count clinically important EEG features will be developed.

SECONDARY OUTCOMES:
Cellular model of developing TSC brain | 2020
  EPIMARKER will develop a innovative human cellular model of epilepsy in developing brain, which can be used for epilepsy biomarkers analyses and for investigations on novel therapeutic strategies in epilepsy.

CONTACTS AND LOCATIONS:
Overall Officials: Sergiusz Jóźwiak, professor, Study Chair — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No